CLINICAL TRIAL: NCT01048242
Title: Treatment of Insomnia in Elderly Sleep Apnea Patients With Ramelteon (TAK 375)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 804640
Record Dates: First submitted 2009-04-15; First posted 2010-01-13 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Insomnia; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea, Obstructive | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramelteon (Experimental): Ramelteon 8 mg oral before bedtime
  Interventions: Drug: rozerem
- sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rozerem — Ramelteon (rozerem) 8mg oral before bedtime
  Other Names: Ramelteon
  Arms: Ramelteon
Drug: Placebo — placebo
  Arms: sugar pill

SUMMARY:
The objective of the study is to determine if treatment with Ramelteon will help to improve insomnia in older adults with co-existent insomnia and sleep apnea. The primary study objective is sleep latency (a measure of insomnia). The hypothesis is that sleep latency will be reduced in subjects taking Ramelteon relative to the placebo arm. The secondary study objective is to determine if subject compliance with CPAP treatment of their sleep apnea is improved in subjects taking Ramelteon (their compliance may be improved because they would have less insomnia due to Ramelteon treatment when using their CPAP). The hypothesis is that compliance with CPAP will be improved in subjects taking Ramelteon relative to the placebo arm.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel arm clinical trial with two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea
* Insomnia
* Age>60

Exclusion Criteria:

* Cognitive impairment
* Active alcohol or substance abuse
* Active use of other sedative-hypnotic agents
* Active use of fluvoxamine (drug interaction with Ramelteon
* Evidence of hepatic dysfunction (Ramelteon contraindicated) on liver function panel
* Presence of Periodic Limb Movement Disorder or Restless Legs Syndrome
* Severe Chronic Obstructive Pulmonary Disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nalaka Gooneratne, MD, MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramelteon | Sugar Pill
Started | 12 | 15
Completed | 8 | 13
Not Completed | 4 | 2
Not completed — See study flow chart | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon | Sugar Pill | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (5.6) | 70.6 (3.5) | 72 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Sleep Onset Latency
Description: Time to sleep onset as determined by polysomnography
Time Frame: 4 weeks
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon | Sugar Pill
Number analyzed (Participants) | 8 | 13
minutes | 9.7 (10.3) | 34.4 (30.7)

ADVERSE EVENTS:
Arm/Group | Ramelteon | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/13
Other Adverse Events (participants affected / at risk) | 4/8 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon (N=8) | Sugar Pill (N=13)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin ulcer--unrelated to study drug treatment, not serious
Paranasal sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Sinusitis--unrelated to study drug treatment, not serious
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Diarrhea--unrelated to study drug treatment, not serious
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Musculoskeletal fracture after being hit by a bicyclist----unrelated to study drug treatment, not serious
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Abdominal pain--unrelated to study drug treatment, not serious
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea--unrelated to study drug treatment, not serious

LIMITATIONS AND CAVEATS:
Auto-Continuous Positive Airway Pressure units used. Single-night of polysomnography Unequal sized arms despite randomization Low rate of completion of at-home sleep diaries Small sample size (pilot study)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No